CLINICAL TRIAL: NCT04587752
Title: Cognitive-Behavioral Therapy for Girls Who Experienced Weight-related Bullying (Online Telehealth Treatment Study)
Brief Title: Cognitive-Behavioral Therapy for Weight-related Bullying (Online Treatment)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000028551
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Bullying; Weight, Body; Trauma, Psychological
Keywords: adolescent; child; cognitive behavioral therapy; eating disorder; obesity
MeSH Terms: conditions — Bullying; Body Weight; Psychological Trauma; Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT for Weight Bullying (Experimental): Cognitive-Behavioral Therapy (CBT) for children who have experienced weight-related bullying
  Interventions: Behavioral: CBT for Weight Bullying

INTERVENTIONS:
Behavioral: CBT for Weight Bullying — Cognitive-behavioral therapy for weight-related bullying delivered by audio/video telehealth.

SUMMARY:
This study will perform a clinical trial with adolescents to pilot a new cognitive-behavioral treatment (CBT) for weight-related bullying testing (1) feasibility, (2) acceptability, and (3) initial efficacy. The treatment will be conducted via audio/video telehealth.

DETAILED DESCRIPTION:
Youth with obesity are more likely to be bullied than healthy-weight peers and weight-related bullying is the most common form of bullying. Treating bullying during childhood could reduce immediate and long-term health consequences, but there are no established individual-level treatments for weight-related bullying despite recommendations that they could improve children's health. This study will develop and test a new treatment for adolescents (11-17 years old) who have experienced bullying due to weight. The treatment will address traumatic stress and potentially co-occurring or developing problems with unhealthy weight-control behaviors, disordered eating, and weight. The treatment will be conducted via audio/video telehealth to increase accessibility and is therefore available to anyone in the United States who meets eligibility criteria.

ELIGIBILITY:
Inclusion Criteria: To be included, adolescents must:

1. Be in the age range ≥11 years old and ≤17 years old;
2. Report experiencing weight-related bullying
3. Report current distress about weight-related bullying
4. Be otherwise-healthy youth (i.e., no uncontrolled or serious medical conditions);
5. Read, comprehend, and write English at a sufficient level to complete study-related materials;
6. Located in the United States and available for participation in the study for 3 months.

Exclusion Criteria: Prospective participants will be excluded if the adolescent:

1. Has a medical or psychiatric condition that would require hospitalization or intensive care (e.g., severe anorexia, neurological disorder, psychotic disorders, suicidality);
2. Has uncontrolled medical condition(s) (e.g., uncontrolled diabetes or hypertension);
3. Is pregnant or breastfeeding;
4. Is taking medication(s) or participating in treatment(s) that could influence weight or appetite;
5. Is engaged in concurrent treatments that focus on trauma-related stress;
6. Began taking hormonal contraceptives less than 3 months prior;
7. Has a developmental or cognitive disorder (e.g., autism spectrum disorder);
8. Has avoidant/restrictive food intake disorder; or
9. Is participating in another clinical research study.

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Identifying as female
Enrollment: 30 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Lydecker, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Lydecker JA, Ozbardakci EV, Lou R, Grilo CM. Trauma-Focused Cognitive-Behavioral Therapy for Adolescents Bullied Because of Weight: A Feasibility Study. Int J Eat Disord. 2024 Oct;57(10):2117-2127. doi: 10.1002/eat.24257. Epub 2024 Jul 15. PMID 39007703

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT for Weight Bullying
Started | 28
Completed | 21
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | CBT for Weight Bullying
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Stress [Mean (Standard Deviation); unit: units on a scale] — Children's Revised Impact of Event Scale (total score; scores range from 0 to 65 with higher scores indicative of more traumatic stress)
  units on a scale | 27.07 (14.20)
Body Dissatisfaction [Mean (Standard Deviation); unit: units on a scale] — Body dissatisfaction subscale of the brief Eating Disorder Examination Questionnaire (weight dissatisfaction and shape dissatisfaction). Population: data not available on two participants.
  units on a scale
    number analyzed (Participants) | 26
    (all) | 3.65 (1.97)
Overvaluation of Shape/Weight [Mean (Standard Deviation); unit: units on a scale] — Overvaluation subscale of the brief Eating Disorder Examination Questionnaire (weight overvaluation and shape overvaluation). Population: data not available on two participants.
  units on a scale
    number analyzed (Participants) | 26
    (all) | 3.37 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Stress
Description: Reductions in traumatic stress as measured by the Children's Revised Impact of Event Scale (total; scores range from 0 to 65 with higher scores indicative of more traumatic stress)
Time Frame: post (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for Weight Bullying
Number analyzed (Participants) | 22
units on a scale | 20.55 (19.07)
Statistical Analysis 1: Comparison: CBT for Weight Bullying; Test type: Superiority; p = .047, t-test, 2 sided

2. Secondary Outcome: Body Dissatisfaction
Description: Reductions in body dissatisfaction (weight and shape dissatisfaction) as measured by the brief Eating Disorder Examination Questionnaire (scores range from 0 to 6; higher scores are indicative of more concern)
Time Frame: post (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for Weight Bullying
Number analyzed (Participants) | 20
units on a scale | 2.85 (2.08)
Statistical Analysis 1: Comparison: CBT for Weight Bullying; Test type: Superiority; p = .01, t-test, 2 sided

3. Secondary Outcome: Overvaluation
Description: Reductions in overvaluation of shape/weight as measured by the brief Eating Disorder Examination Questionnaire (scores range from 0 to 6; higher scores are indicative of more concern)
Time Frame: post (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for Weight Bullying
Number analyzed (Participants) | 20
units on a scale | 1.93 (1.83)
Statistical Analysis 1: Comparison: CBT for Weight Bullying; Test type: Superiority; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CBT for Weight Bullying
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04587752/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04587752/ICF_001.pdf